CLINICAL TRIAL: NCT00201123
Title: Host Response to Tuberculosis and Acquired Immune Deficiency Syndrome
Brief Title: Effects of Interferon-Gamma on Cavitary Pulmonary Tuberculosis in the Lungs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 264; R01HL059832-06 (NIH)
Record Dates: First submitted 2005-09-16; First posted 2005-09-20 (Estimated); Results first posted 2014-06-10 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Tuberculosis; AIDS-related Complex
MeSH Terms: conditions — Tuberculosis; AIDS-Related Complex

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard Treatment (Placebo Comparator): Isoniazid, Rifampin, Pyrazinamide Anti-Tuberculous Therapy
  Interventions: Other: Placebo
- Aerosol Interferon-gamma (Experimental): Aerosol Interferon-Gamma plus Isoniazid, Rifampin, and Pyrazinamide
  Interventions: Drug: Aerosol Interferon-Gamma
- Subcutaneous Interferon-Gamma (Experimental): Subcutaneous Interferon-Gamma plus Isoniazid, Rifampin, and Pyrazinamide
  Interventions: Drug: Subcutaneous interferon-gamma

INTERVENTIONS:
Drug: Aerosol Interferon-Gamma — Participants will receive aerosol interferon-gamma.
  Arms: Aerosol Interferon-gamma
Drug: Subcutaneous interferon-gamma — Patients will receive subcutaneous interferon-gamma
  Arms: Subcutaneous Interferon-Gamma
Other: Placebo
  Arms: Standard Treatment

SUMMARY:
This study will evaluate the lung's immune response to mycobacterium tuberculosis (Mtb) infection and will modulate that response with interferon-gamma.

DETAILED DESCRIPTION:
BACKGROUND:

Mtb infects one-third of the world's population and ranks seventh in terms of global morbidity and mortality. Patients with bilateral pulmonary tuberculosis (TB), cavitary disease, and persistently positive sputum smears pose a special risk for treatment failure and/or relapse.

DESIGN NARRATIVE:

Cavitary pulmonary TB will be studied and interferon-gamma will be used as the intervention. The outcome of this study will be the changes in mycobacteriology, chest radiography, and bronchoalveolar lavage (BAL) cells.

The primary outcome will be sputum conversion, which will be measured at Weeks 4 and 8.

The key secondary outcomes of this study will include a chest computerized tomography (CT) scan and BAL to measure the flow of cytometry and cytokine levels. Both outcomes will be measured at baseline and at Month 4.

ELIGIBILITY:
Inclusion Criteria:

* Positive acid-fast bacillus (AFB) smear within 14 days prior to randomization
* Cluster of Differentiation 4 greater than 200 if HIV positive
* Ability to sign consent
* Bilateral, cavitary pulmonary TB

Exclusion Criteria:

* Multidrug-resistant (MDR) TB
* Extrapulmonary TB
* HIV positive with opportunistic infection within 30 days of study entry
* Cancer
* Asthma
* Pregnant or lactating women
* Chronic heart disease
* Chronic liver disease
* Chronic renal disease
* Seizure disorder
* Bleeding or clotting disorder
* Diabetes mellitus

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2005-04; Primary Completion 2007-01 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Rom, MD, MPH, Principal Investigator — NYU School of Medicine
Locations (2):
- NYU School of Medicine, New York, New York, United States
- The Lung Institute at University of Cape Town, Cape Town, South Africa

REFERENCES:
- [Result] Dawson R, Condos R, Tse D, Huie ML, Ress S, Tseng CH, Brauns C, Weiden M, Hoshino Y, Bateman E, Rom WN. Immunomodulation with recombinant interferon-gamma1b in pulmonary tuberculosis. PLoS One. 2009 Sep 15;4(9):e6984. doi: 10.1371/journal.pone.0006984. PMID 19753300

RESULTS

PARTICIPANT FLOW:
Groups:
- DOTS Control Group: DOTS Control Group
  IRPE Anti-Tuberculous Therapy: Participants will receive IRPE anti-tuberculous therapy.
- Aerosol Interferon Gamma for TB: Aerosol Interferon-Gamma
  Aerosol Interferon-Gamma: Participants will receive aerosol interferon-gamma.
- Subcutaneous Interferon Gamma for TB: Subcutaneous Interferon-Gamma
  Subcutaneous Interferon-Gamma: Partcipants will receive subcutaneous interferon-gamma.
Period: Overall Study
Arm/Group | DOTS Control Group | Aerosol Interferon Gamma for TB | Subcutaneous Interferon Gamma for TB
Started | 32 | 32 | 32
Did Not Meet Continuation Criteria | 2 | 0 | 5
Completed | 26 | 28 | 23
Not Completed | 6 | 4 | 9

BASELINE CHARACTERISTICS:
Population: Demographic information provided for all subjects who were eligible for the study after all screening procedures were performed. 7 subjects who were found to be ineligible after randomization but prior to administration of treatment (listed as "did not meet continuation criteria" in participant flow section) are not included in baseline analysis.
Groups:
- DOTS Control Group: IRPE Anti-Tuberculous Therapy
  IRPE Anti-Tuberculous Therapy: Participants will receive IRPE anti-tuberculous therapy.
- Subcutaneous Interferon Gamma for TB: Subcutaneous Interferon-Gamma
  Subcutaneous Interferon-Gamma: Participants will receive subcutaneous interferon-gamma.
- Total: Total of all reporting groups
Arm/Group | DOTS Control Group | Aerosol Interferon Gamma for TB | Subcutaneous Interferon Gamma for TB | Total
Number analyzed (Participants) | 30 | 32 | 27 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (11) | 34 (10) | 35 (13) | 34 (10)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 32 | 27 | 89
  >=65 years | 0 | 0 | 0 | 0
Gender [Count of Participants; unit: Participants]
  Female | 10 | 8 | 9 | 27
  Male | 20 | 24 | 18 | 62
Region of Enrollment [Number; unit: participants]
  South Africa | 30 | 32 | 27 | 89

OUTCOME MEASURES:

1. Primary Outcome: Sputum Conversion
Time Frame: Measured at 16 Weeks
Population: Intention to Treat analysis performed. Only subjects excluded were those who did not receive treatment.
Measure: Number; unit: percentage of participants
Arm/Group | DOTS Control Group | Aerosol Interferon Gamma for TB | Subcutaneous Interferon Gamma for TB
Number analyzed (Participants) | 30 | 32 | 27
percentage of participants | 36 | 60 | 36

2. Secondary Outcome: Chest Cavity Size
Time Frame: 16 Weeks
Population: Intention to Treat analysis performed. Only subjects excluded were those who did not receive treatment.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | DOTS Control Group | Aerosol Interferon Gamma for TB | Subcutaneous Interferon Gamma for TB
Number analyzed (Participants) | 32 | 30 | 27
millimeters
  Baseline | 34 (11) | 39 (24) | 34 (13)
  16 Weeks | 20 (16) | 29 (24) | 18 (17)

3. Secondary Outcome: Bronchoalveolar Lavage (BAL) to Measure Flow of Cytometry and Cytokine Levels
Time Frame: 16 Weeks
Population: Intention to Treat analysis performed. Only subjects excluded were those who did not receive treatment.
Measure: Median (Inter-Quartile Range); unit: cells/mL
Arm/Group | DOTS | Nebulized rlFN-y | Subcutaneous rlFN-y
Number analyzed (Participants) | 30 | 32 | 27
cells/mL
  Lymphocytes Week 0 | 4 [2 to 8] | 5 [3 to 15] | 6 [3 to 10]
  Lymphocytes Week 16 | 15 [6 to 25] | 15 [8 to 34] | 22 [13 to 33]
  Machrophages Week 0 | 60 [17 to 84] | 60 [32 to 80] | 62 [43 to 83]
  Machrophages Week 16 | 64 [44 to 72] | 63 [40 to 84] | 66 [54 to 77]
  Neutrophils Week 0 | 28 [10 to 82] | 24 [5 to 56] | 30 [4 to 54]
  Neutrophils Week 16 | 11 [3 to 31] | 4 [2 to 16] | 2 [2 to 9]

ADVERSE EVENTS:
Arm/Group | DOTS Control Group | Aerosol Interferon Gamma for TB | Subcutaneous Interferon Gamma for TB
Serious Adverse Events (participants affected / at risk) | 1/30 | 3/32 | 3/27
Other Adverse Events (participants affected / at risk) | 0/30 | 0/32 | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DOTS Control Group (N=30) | Aerosol Interferon Gamma for TB (N=32) | Subcutaneous Interferon Gamma for TB (N=27)
hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Desaturation on BAL (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No